CLINICAL TRIAL: NCT02192281
Title: Randomized Experiment of Playworks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MPR-06758; 12-177 (Other: New England Institutional Review Board)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Focus on Physical Activity, Recess, and Play
Keywords: Physical activity; Recess; Accelerometer; Play
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Playworks (Experimental): Playworks was implemented during the entire school year, and outcome measures were collected in spring of the school year.
  Interventions: Other: Playworks
- Control (No Intervention): Playworks was not implemented at these schools.

INTERVENTIONS:
Other: Playworks — The Playworks program places full-time coaches in low-income schools to provide opportunities for organized play during recess and throughout the school day.
  Arms: Playworks

SUMMARY:
The purpose of this study is to determine whether Playworks has an impact on student and school outcomes such as physical activity, behavior, and academic performance.

DETAILED DESCRIPTION:
Playworks is a school-based program that places full-time coaches in low-income schools to organize games and activities during recess. The Robert Wood Johnson Foundation (RWJF) contracted with Mathematica Policy Research and its subcontractor, the John W. Gardner Center for Youth and Their Communities (JGC) at Stanford University, to conduct a rigorous evaluation of Playworks. Twenty-nine schools interested in implementing Playworks, across six cities in the United States, were randomly assigned to treatment and control groups during the 2010-2011 (cohort 1) or 2011-2012 (cohort 2) school year. Random assignment was conducted within matched groups of schools within each city. In total, there were 12 blocks of matched schools. For each block, one school was randomly assigned to the control group and the rest to the treatment group.

During the one-year study period for each cohort, treatment schools received Playworks and control schools were not eligible to implement Playworks. Data from student surveys, accelerometers, and teacher surveys were collected from 4th- and 5th-grade students, teachers, and school staff roughly seven months after Playworks was first implemented in treatment schools.

For the student survey, students were asked to complete a 30-minute student survey in the spring of their study year about their experiences at school. A team of experienced survey administration staff administered the survey in the students' classrooms. In addition to the student survey, teachers were asked to complete a teacher survey that asked teachers about their students' experiences at school.

A subsample of students that were asked to complete the student survey also wore accelerometers during one or two school days. During the accelerometer data collection period, the research team arrived at participating classrooms at the beginning of the school day. Team members described the function of the accelerometer and then attached one to each consented student's hip, using an elastic belt. The accelerometer data was then processed with the ActiLife 5 software package.

The impact of Playworks on study outcomes was estimated by comparing the average outcomes in treatment and control schools using regression models customized to the unit of analysis (teacher or student). The regression models used for analysis included indicators for random assignment blocks to account for the blocked design and school-specific random error terms to account for school-specific effects not attributable to the treatment. Covariates were also included in some models to account for significant differences between treatment and control groups in demographic characteristics. Models for continuous and binary outcome variables were fit using least-squares estimation and logistic regression estimation, respectively. Standard errors for the estimated impacts on teacher- and student-level outcomes accounted for clustering at the school level using generalized estimating equations. Model-based p-values and effect sizes were calculated based on the estimated impacts and corresponding standard errors and multiple comparison adjustments accounted for correlations among the multiple tests. Sampling weights were used when estimating impacts. The weights were constructed to account for both the selection probabilities of students and teachers into the sample and nonresponse.

ELIGIBILITY:
Inclusion Criteria:

* Students in low-income schools in urban areas
* Students in schools where at least 50 percent of students qualify for free or reduced-price lunch.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2278 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Mean Number of Accelerometer Intensity Counts Recorded Per Minute During Recess | 8 weeks
Mean Number of Steps Taken Per Minute During Recess | 8 weeks
Mean Percentage of Accelerometer Wear Time During Recess Spent in Sedentary Activity | 8 weeks
Mean Percentage of Accelerometer Wear Time During Recess Spent in Light Activity | 8 weeks
Mean Percentage of Accelerometer Wear Time During Recess Spent in Moderately Intense Activity | 8 weeks
Mean Percentage of Accelerometer Wear Time During Recess Spent in Vigorously Intense Activity | 8 weeks

SECONDARY OUTCOMES:
Percentage of Students Who Participate in Recess Activities That Make Them Sweat and Breathe Hard "Sometimes" or "A Lot" | 8 weeks
Percentage of Teachers Who "Agree" or "Strongly Agree" That Their Students Participate in Physical Activities That Make Them Sweat and Breathe Hard During Recess | 8 weeks
Percentage of Students Who Participated in a Sports Team After School or on the Weekend During the School Year | 8 weeks
Percentage of Students Who Participated in Dance, Gymnastics or Martial Arts Lessons After School or on the Weekend During the School Year | 8 weeks

OTHER OUTCOMES:
Participation in Individual Activities During Recess Scale Score | 8 weeks
Participation in Games During Recess Scale Score | 8 weeks
Percentage of Students Who Report That the Following Happens "Sometimes" or "A Lot": Adults help them play games and sports during recess | 8 weeks
Percentage of Students Who Report That the Following Happens "Sometimes" or "A Lot": Their teacher helps them play games and sports during recess | 8 weeks
Percentage of Students Who Report That the Following Happens "Sometimes" or "A Lot": They talk with friends during recess | 8 weeks
Recess Behavior and Readiness for Class Scale Score | 8 weeks
Recess Misbehavior/Discipline Scale Score | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Ask an adult to help them solve a conflict during recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Get teased about not being good at games or sports during recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Get into an argument with other students during recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Fight or hit other students during recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Work out problems with other students during recess without fighting | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Say encouraging things to other students during recess | 8 weeks
Enjoyment of Recess Scale Score | 8 weeks
Percentage of Students Who Agree "A Little" or "A Lot" That They: Like to play games and sports at recess | 8 weeks
Percentage of Students Who Agree "A Little" or "A Lot" That They: Feel like they can join other kids in a game on the playground | 8 weeks
Percentage of Students Who Agree "A Little" or "A Lot" That They: Feel left out at recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Get to play a game that they want during recess | 8 weeks
Percentage of Students Who Report That They Do the Following "Sometimes" or "A Lot": Have to play a game that adults want them to play during recess | 8 weeks
Games and Sports Self-Concept Scale Score | 8 weeks
Percentage of Teachers Who "Agree" or "Strongly Agree" That Their Students: Look forward to recess | 8 weeks
Percentage of Teachers Who "Agree" or "Strongly Agree" That Their Students: Enjoy adult-organized activities at recess | 8 weeks
Percentage of Teachers Who "Agree" or "Strongly Agree" That Their Students: Would be upset about missing recess | 8 weeks
Percentage of Teachers Who "Agree" or "Strongly Agree" That Their Students: Feel ownership over their activities during recess | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne James-Burdumy, Principal Investigator — Mathematica Policy Research; Martha Bleeker, Study Director — Mathematica Policy Research
Locations (1):
- Mathematica Policy Research, Princeton, New Jersey, United States